CLINICAL TRIAL: NCT05154084
Title: Transurethral REsection and Single Instillation Intra-vesical Chemotherapy Evaluation in Bladder Cancer Treatment (RESECT) Improving Quality in TURBT Surgery
Brief Title: RESECT: Improving Quality in TURBT Surgery.
Acronym: RESECT
Status: Completed | Type: Observational
Sponsor: British Urology Researchers in Surgical Training (Other)
Collaborators: Action Bladder Cancer UK (Other); British Journal of Urology International (Unknown); Rosetrees Trust (Other); Photocure (Industry); KARL STORZ Endoscopy-America, Inc. (Industry); University College, London (Other); University of Aberdeen (Other); The Urology Foundation, United Kingdom (Unknown)
Responsible Party: Sponsor
Other Study IDs: RESECT Protocol 4.0 111120
Record Dates: First submitted 2021-10-29; First posted 2021-12-10 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Bladder Cancer
Keywords: Non muscle-invasive bladder cancer; Urothelial carcinoma; Collaborative study; Quality improvement
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms; Carcinoma, Transitional Cell | interventions — Educational Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Audit only: This group of sites will participate in the audit. No performance feedback will be provided during the period under study. Feedback will be provided at the end of the study period.
- Audit with feedback: This group of sites will participate in the audit, and receive a feedback intervention about their practice based on retrospective data about surgery performed before the start of the study period.
  Interventions: Behavioral: Performance feedback and education

INTERVENTIONS:
Behavioral: Performance feedback and education — Hospitals and surgeons will have an online interactive performance feedback dashboard provided to them along with educational components.
  Groups: Audit with feedback

SUMMARY:
Superficial bladder cancer, known as non-muscle-invasive bladder cancer (NMIBC), is the most common type of bladder cancer. It is expensive to manage and significantly impacts on patients' quality of life. This is because there is a high burden of recurrent disease after initial treatment, and need for long term surveillance for recurrence.

The most important step in the diagnosis and treatment of NMIBC is the first surgical procedure called the transurethral resection of bladder tumour (TURBT). There is evidence that the quality of the TURBT operation, and the use of a single administration of bladder chemotherapy following the operation, can reduce cancer recurrence rates and progression to more invasive cancer. There is anecdotal evidence that the quality of TURBT surgery and the usage of intravesical chemotherapy varies widely between hospitals and thus may result in worse outcomes for some patients.

The primary objective of the study is to determine if audit and feedback can improve the quality of TURBT surgery and if this reduces recurrence of NMIBC.

DETAILED DESCRIPTION:
RESECT aims to be the largest multicentre international observational study evaluating the first and most important step in the management of non muscle-invasive bladder cancer (NMIBC), the transurethral resection of bladder tumour (TURBT).

It is known that achieving a "good quality" TURBT results in reduced NMIBC recurrence rates. This evidence forms the basis for the recommendations made in evidence-based guidelines such as the European Association of Urology (EAU), the American Urological Association (AUA) and the National Institute for Health and Care Excellence (NICE). The RESECT study will evaluate the effects of a variety of patient, hospital, surgical and surgeon-related factors which may contribute to altered outcome in patients with NMIBC following a TURBT.

The only known national data collection about quality standards in TURBT surgery is in Scotland. The aim is to conduct a multicentre international observational study of urological practice for the management of NMIBC. Current operative practice will be measured across hospitals, regions and countries and compare these against evidence-based recommendations. It will be determined if any hospital, service, training or technical factors impact the achievement of quality indicators and/or early recurrence rates. These data will be used to present hospital and surgeon performance back to surgeons as an intervention to drive quality improvement. The timing of feedback to different hospitals will be varied randomly so that it can determined if the feedback is having an impact on audit performance.

RESECT aims to answer some key UNKNOWNS:

Does reporting and comparing our TURBT quality make us do it better? What things should be measured to determine TURBT quality? What rate of achievement should be aimed for in our practice? What factors are associated with better achievement of TURBT quality?

Methods:

The is an observational study that will include randomized feedback and education to hospitals about their TURBT performance.

Sites will first submit survey data about usual practice, and then retrospective data about consecutive TURBT surgery previously performed at their site.

Sites will then be randomized to either receiving early feedback or to not receiving early feedback and just taking part in the study. Sites will then collect prospective data about consecutive TURBT surgeries performed at their site.

Performance will then be compared between hospitals that received feedback during the study and those who did not. All sites will receive the feedback intervention at the end of the study.

ELIGIBILITY:
Site inclusion criteria:

Perform TURBT surgery for non-muscle invasive bladder cancer and perform at least 20 first tumour TURBT surgeries per year.

Case Inclusion criteria:

● Patients undergoing transurethral surgical treatment of confirmed transitional cell carcinoma of the bladder

Case Exclusion criteria

* Radiologically suspected muscle invasive bladder cancer pre-operatively
* Surgery not performed with curative intent: a. Diagnostic purposes only b. Symptomatic or palliative purposes only c. diffuse lesions that cannot cured by TURBT surgery
* Emergency TURBT
* Records lacking pre-defined minimum data set
* All records from sites where the study minimum requirements are not met

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Site: Primary analysis and randomization is at the site level. Patients are not randomized and audit performance outcomes are analysed at the site level. Estimated 200 sites total sample.
  Patient: Patients undergoing TURBT for a first or recurrent transitional cell carcinoma presumed to be non-muscle invasive at the time of surgery.
Sampling Method: Non-Probability Sample
Enrollment: 19505 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
The rate of detrusor muscle sampling at TURBT | At point of surgery, assessed from specimen pathology report.
  The proportion of first tumour cases with tumours >5mm in diameter where detrusor muscle is present in the specimen on histological assessment.
The rate of single instillation intra-vesical chemotherapy (SI-IVC) instillation within 24 hours | 24 hours.
  The proportion of first tumour cases at sites where SI-IVC is possible that were given SI-IVC within 24 hours of TURBT.
The rate of documentation of resection completeness | At time of surgery, assessed retrospectively from patient record.
  The proportion of first tumour cases where a statement of resection completeness is included in the patient operation record.
The rate of documentation of all of tumour number, tumour size and tumour location in the operative record. | At time of surgery, assessed retrospectively from patient record.
  The proportion of first tumour cases where all of tumour number, tumour size and tumour location are documented in the official operative record.

SECONDARY OUTCOMES:
Early recurrence rate | 12 months
  The rate of recurrence at first follow up check after complete TURBT.
The rate of achievement of all applicable key TURBT quality indicators | 12 months
  The proportion of first tumour cases achieving all applicable co-primary outcomes. This is a composite outcome that aims to determine if a single metric of quality is associated with cancer recurrence.
The rate of Clavien Dindo 3 or more complications | 1 month after surgery
  The rate of Clavien Dindo 3 or more complications
The association of the achievement of TURBT quality indicators with early recurrence. | 12 months.
  A per protocol and per-protocol analysis will be performed to determine if actual achievement of TURBT quality indicators is association with early recurrence rate.
The association of en-bloc resection or use of visual diagnostic aids with achievement of TURBT quality indicators and early recurrence rate | 12 months
  To determine if the use of en-bloc resection or visual diagnostic aids improves achievement of quality indicators and reduces recurrence
The association of surgeon experience in years and number of TURBTs performed per month with achievement of TURBT quality indicators and early recurrence rate | 12 months
  To determine if surgical experience is important in TURBT quality
The association of dedicated TURBT lists with achievement of TURBT quality indicators and early recurrence rate | 12 months
  To determine if focusing one type of surgery (TURBT) in a dedicated surgical list improves outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Veeru Kasivisvanathan, MBBS, Principal Investigator — University College, London
Locations (1):
- BURST, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Country specific data to be provided to regional lead on request and with conditions.

REFERENCES:
- [Derived] Gallagher K, Bhatt N, Clement K, Zimmermann E, Khadhouri S, MacLennan S, Kulkarni M, Gaba F, Anbarasan T, Asif A, Light A, Ng A, Chan V, Nathan A, Cooper D, Aucott L, Marcq G, Teoh JY, Hensley P, Duncan E, Goulao B, O'Brien T, Nielsen M, Mariappan P, Kasivisvanathan V. Audit, Feedback, and Education to Improve Quality and Outcomes in Transurethral Resection and Single-Instillation Intravesical Chemotherapy for Nonmuscle Invasive Bladder Cancer Treatment: Protocol for a Multicenter International Observational Study With an Embedded Cluster Randomized Trial. JMIR Res Protoc. 2023 Jun 15;12:e42254. doi: 10.2196/42254. PMID 37318875